CLINICAL TRIAL: NCT02798887
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of Membrane vs. no Membrane Approach to Grafting.
Brief Title: Ridge Preservation Comparing the Healing With or Without a Barrier Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.0461
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Regeneration; Bone regeneration; Grafting, Bone; Allograft; Xenograft
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ridge preservation membrane (Experimental): Positive control Patients will receive ridge preservation intrasocket allograft and overlay xenograft resorbable with membrane
  Interventions: Procedure: Ridge preservation
- Ridge preservation no membrane (Experimental): test patients will receive ridge preservation intrasocket allograft and overlay xenograft with no membrane
  Interventions: Procedure: Ridge preservation

INTERVENTIONS:
Procedure: Ridge preservation — Ridge preservation comparing the clinical and histologic healing with or without a barrier membrane

SUMMARY:
Ridge Preservation Comparing the Clinical and Histologic Healing of Membrane vs. no Membrane Approach to Grafting.

DETAILED DESCRIPTION:
Thirty patients will be treated using the principles of bone grafting for ridge preservation. Fifteen test patients will receive a flap technique with an intrasocket cancellous cortical particulate allograft plus a facial overlay graft using a bovine xenograft without a membrane where only the exposed intrasocket allograft will be covered with a piece of Alloderm GBR. The positive control group of fifteen patients will receive a flap technique with an intrasocket cancellous cortical particulate allograft plus a facial overlay graft using a bovine xenograft plus Alloderm GBR membrane. Approximately, four months post-surgery, a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Change in post-extraction site to 4 month change in crestal osseous width | 4 months
  Changes in post-extraction to 4 month change in ridge measurements at the mid defect alveolar crest and 5 mm apical taken with a caliper.

SECONDARY OUTCOMES:
Change in Soft tissue thickness | 4 months
  Soft tissue thickness measurements taken with a #40 endodontic reamer.
Percent osseous tissue | 4 months
  A trephine core will be harvested at 4 months. Following histologic processing the osseous core will be classified into percent vital bone, nonvital bone and trabecular space.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MSD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic University of Louisville, Louisville, Kentucky, United States